CLINICAL TRIAL: NCT01277224
Title: Effectiveness of a Leisure Time Physical Activity Intervention on the Overweight and the Obesity in Schoolchildren. The Cuenca's Study
Brief Title: Effectiveness of a Physical Activity Intervention on the Obesity of Schoolchildren
Acronym: Movi2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, FRANCISCO QUILES VICECHANCELLOR OF RESEARCH, Proffesor, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI081297
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Physical Activity; Obesity; Children
Keywords: physical activity; obesity; adiposity; children; blood lipids; blood pressure; randomized controlled trials
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Movi2 Program (Experimental)
  Interventions: Behavioral: Movi2 Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Movi2 Program — In the Movi2 program we will perform a recreational physical activity intervention during one year that include standardized recreative and non competitive activities conducted by sports instructors. It consisted of two 90-min after school sessions per week on school days and one 150-minute session on Saturday morning.
  Arms: Movi2 Program

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a recreational physical activity intervention (RPAI) for reducing the prevalence of overweight/obesity and other cardiovascular risk factors

DETAILED DESCRIPTION:
The prevalence of overweight in Spanish children in the puberty age is among the highest in the world and increasing quickly. The investigators recently evaluated an after-school program of recreational physical activity to control obesity and other cardiovascular risk factors in primary school children in Cuenca. This program, known as the Movi program, reduced adiposity, increased serum apolipoprotein (apo) A-I concentration and reduced apo B concentration over one-year period.

Though the intervention MOVI had great acceptance between the children and his families, and it demonstrated to be effective opposite to the obesity, his results were relatively modest. For it, our hypothesis of work, which justifies this new project, is that a major intensity of the intervention, and a major weekly duration extending this one to the weekend, it might improve the efficiency on the obesity.

ELIGIBILITY:
The Boards of Governors (community participatory organ in each school) and the children's parents will inform of the study's aims and methods, and give their written consent to the children's participation. Similarly, the study will present classroom-by-classroom to the children, and their oral consent will obtain. Participant children will be free of serious learning difficulties, or physical or mental disorders, that could impede participation in the scheduled physical activities.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Skin-fold thickness | 1 year
  Over 1 years, the Movi program will reduce the prevalence of excess weight in schoolchildren and improve other cardiovascular risk factors.

SECONDARY OUTCOMES:
Physical activity, physical fitness, sleep, and quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Martinez-Vizcaíno, PhD, Principal Investigator — Health and Social Research Centre, Universidad de Castilla-La Mancha, Cuenca, Spain

REFERENCES:
- [Derived] Nystrom CD, Henriksson P, Martinez-Vizcaino V, Medrano M, Cadenas-Sanchez C, Arias-Palencia NM, Lof M, Ruiz JR, Labayen I, Sanchez-Lopez M, Ortega FB. Does Cardiorespiratory Fitness Attenuate the Adverse Effects of Severe/Morbid Obesity on Cardiometabolic Risk and Insulin Resistance in Children? A Pooled Analysis. Diabetes Care. 2017 Nov;40(11):1580-1587. doi: 10.2337/dc17-1334. Epub 2017 Sep 22. PMID 28939688
- [Derived] Martinez-Vizcaino V, Sanchez-Lopez M, Notario-Pacheco B, Salcedo-Aguilar F, Solera-Martinez M, Franquelo-Morales P, Lopez-Martinez S, Garcia-Prieto JC, Arias-Palencia N, Torrijos-Nino C, Mora-Rodriguez R, Rodriguez-Artalejo F. Gender differences on effectiveness of a school-based physical activity intervention for reducing cardiometabolic risk: a cluster randomized trial. Int J Behav Nutr Phys Act. 2014 Dec 10;11:154. doi: 10.1186/s12966-014-0154-4. PMID 25491026
- [Derived] Martinez-Vizcaino V, Sanchez-Lopez M, Salcedo-Aguilar F, Notario-Pacheco B, Solera-Martinez M, Moya-Martinez P, Franquelo-Morales P, Lopez-Martinez S, Rodriguez-Artalejo F; MOVI-2 group. Protocol of a randomized cluster trial to assess the effectiveness of the MOVI-2 program on overweight prevention in schoolchildren. Rev Esp Cardiol (Engl Ed). 2012 May;65(5):427-33. doi: 10.1016/j.recesp.2011.12.008. Epub 2012 Mar 10. English, Spanish. PMID 22410389